CLINICAL TRIAL: NCT05743114
Title: Non-Invasive, Non-pharmacologic, Computer Interface Approach to Modulate Electroencephalogram (EEG) Potentials, Alertness and Sleep With Acoustic Stimulation
Brief Title: Sounds Locked to ElectroEncephalogram Phase For the Acceleration of Sleep Onset Time
Acronym: SLEEPFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elemind Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-02-13
Record Dates: First submitted 2023-02-06; First posted 2023-02-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Sleep; Sleep Disturbance
Keywords: Neuromodulation; Electroencephalogram; Auditory Stimulation; Sleep; Wake After Sleep Onset
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Conditions are blinded to the participant and during data analysis and sleep scoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Onset Latency Crossover (Experimental): Arm 1 is a crossover arm in which participants receive one block of active stimulation (experimental) and a second block in which the device is worn and actively recording, but not delivering phase-locked auditory stimulation (sham). The order of blocks is randomized for each participant.
  Interventions: Device: Elemind Neuromodulation (ENMod)
- Wake After Sleep Onset (Experimental): This arm tests active stimulation during sleep onset, as well as additional stimulation if participants wake up during the night. One of 4 possible conditions are randomized for each stimulation even (within subject and within nights): Stimulation locked to alpha peak phase, stimulation locked to alpha trough phase, white noise (active sham), and no sound (control).
  Interventions: Device: Elemind Neuromodulation (ENMod)

INTERVENTIONS:
Device: Elemind Neuromodulation (ENMod) — The ENMod is a headband that measures electroencephalogram (EEG) activity, computes the phase of neural oscillations in real-time, and delivers auditory pulses intended to interact with ongoing neural oscillations.

SUMMARY:
This study seeks to test whether auditory stimulation delivered at specific phases of the alpha oscillation (as measured by electroencephalogram) can accelerate sleep onset.

DETAILED DESCRIPTION:
In healthy sleepers, cortical alpha oscillations are present during the transition from wakefulness to sleep, and dissipate at sleep onset. For individuals with insomnia, alpha power is elevated during the wake-sleep transition and can persist throughout the night. This study tests whether a wearable device that delivers auditory stimulation phase-locked to alpha oscillations can accelerate sleep onset in healthy adults who report difficulties falling and staying asleep. The device is a prototype of the Elemind Neuromodulation system (ENMod). The ENMod is a wireless headband that measures brain signals, computes the phase of neural oscillations in specific frequency bands, and delivers audible pink noise pulses at specific times relative to the instantaneous phase of neural oscillations. In this study, we ask participants to wear the ENMod headband at home while going to sleep. The device is programmed to record EEG activity and, during the transition from wakefulness to sleep, deliver phase-locked sounds that are intended to interact with the participants neural activity and accelerate sleep onset.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent after reading and answering questions in written English
* Self-report that it takes 30 minutes on average or more to fall asleep
* Subthreshold to Moderately severe Clinical insomnia symptoms (ISI < 21)
* Subthreshold to Moderately severe Clinical insomnia (PSQI > 6)
* Minimal risk for severe Generalized Anxiety Disorder (GAD-7 < 15)
* Minimal risk for severe Generalized Anxiety Disorder (GAD-7 < 15)
* Individuals that are not actively being treated for anxiety, insomnia, ADHD or other psychological disorders with medications
* Self-report of difficulty staying asleep "Moderate," "Severe," or "Very Severe"
* Self report of waking up in the middle of the night/early morning one or more times per week

Exclusion Criteria:

* Unable to read or understand English
* Body Mass Index (weight/height ratio) >33
* Self-report of being diagnosed with apnea
* Current or past history of a neurological disorder or psychiatric illness
* Self-report that it takes less than 30 minutes to fall asleep on average
* Severe Clinical insomnia symptoms (ISI > 21)
* Good sleepers (PSQI < 6)
* High risk for severe Generalized Anxiety Disorder (GAD-7 > 15)
* Moderate to high risk for alcohol abuse disorder (AUDIT >6)
* individuals that are actively being treated for anxiety, insomnia, ADHD or other psychological disorders with medications
* Consumption of more than 4 cups of Caffeinated beverages per day
* Any caffeine < 6hrs prior to each recording session (e.g. coffee, tea, caffeinated sodas etc.)
* Any seizures or family history of seizures
* History of migraine
* History of brain related injury or unexplained loss of consciousness
* Cardiac pacemaker or intracranial metal implant
* Pregnant
* Taking any anti-depressants, stimulants, medication for hypertension or hypotension and/or cannabis derived products
* Cochlear implant in either ear
* Diagnosed with hearing impairment or deafness
* Works night shifts any night of the week

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Onset Latency (SOL) from Sham Block Compared to Stimulation Block | At the completion of the study (14 days), including at least 4 days in each block.
  SOL will be determined using objective EEG-based metrics (e.x. time to first observed sleep spindle) derived from recommendations set forth by the American Academy of Sleep Medicine (AASM). SOL will be assessed for each study day during the sham block in which the device is worn but inactive and compared to SOL for the days in the stimulation block, in which the device is actively delivering auditory stimulation. Subjects will randomly be assigned in regards to the order of sham and stimulation blocks.

SECONDARY OUTCOMES:
Change in Sleep Efficiency During Sham Block Compared to Stimulation Block | At the completion of the study (14 days), including at least 4 days in each block.
  Sleep efficiency, defined as the percentage of time spent asleep out of the total time spent in bed will assessed for each study day during the sham block in which the device is worn but inactive and compared to the sleep efficiency for each day in the stimulation block, in which the device is actively delivering auditory stimulation. Subjects will randomly be assigned in regards to the order of sham and stimulation blocks.
Sleep Onset Latency After Wake After Sleep Onset Events (WASO) During Sham Stimulation Sessions Compared to Active Stimulation Sessions | At the completion of the study (7-14 days).
  Sleep onset latency will be measured after middle-of-night wake up events using EEG-based metrics according to guidelines set forth by the American Academy of Sleep Medicine (AASM). Stimulation condition (sham or active) will be randomized for each WASO event (including events within a single night as well as across all nights). At the completion of the study, SOL will be compared for WASO events in which sham stimulation was delivered compared to WASO events in which active stimulation was delivered.
Change in Subjective Sleep Onset Latency (SOL) from Sham Block Compared to Stimulation Block | At the completion of the study (14 days).
  Subject-reported time to fall asleep will be assessed using the results from a questionnaire that includes the first 9 questions from the Consensus Sleep Diary (Carney et al., 2012). This survey asks the participant to report bed time, wake time, the amount of time it took to fall asleep, the number of awakenings during the night and the total duration of such awakenings. The questionnaire also asks the subject to rate quality of sleep on a 5-point scale from very poor to very good. The reported time to fall asleep on days during the sham block will be compared to the same metric reported on days during the stimulation block.
Change in Subjective Daytime Sleepiness (Karolinska Sleepiness Scale) from Sham Block Compared to Stimulation Block | At the completion of the study (14 days).
  Subject-reported feelings of sleepiness and alertness during the day will be assessed using the Karolinska Sleepiness Scale (KSS) questionnaire. This is a single question scale on which sleepiness is assessed using a score from 1-9, with 1 representing a level of high alertness, and 9 representing very sleepy. The reported KSS score during the sham block will be compared to the same metric reported on days during the stimulation block.

CONTACTS AND LOCATIONS:
Locations (1):
- Elemind Technologies, Inc, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Derived] Bressler S, Neely R, Yost RM, Wang D. A randomized controlled trial of alpha phase-locked auditory stimulation to treat symptoms of sleep onset insomnia. Sci Rep. 2024 Jun 6;14(1):13039. doi: 10.1038/s41598-024-63385-1. PMID 38844793